CLINICAL TRIAL: NCT07126301
Title: Assessing the Feasibility of Aromatherapy Essential Oil Associated Changes on Nausea in Patients Receiving Infusion in the Ambulatory Setting
Brief Title: Aromatherapy Essential Oils to Manage Anxiety and Nausea in Cancer Patients Receiving Infusion in the Ambulatory Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24459; NCI-2025-04956 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24459 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-07-28; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm I (peppermint oil) (Experimental): Patients inhale peppermint essential oil via the PID once every hour starting on day 1 during their anti-cancer/chemotherapy infusions. Patients continue to inhale the peppermint essential oil via the PID at least three times a day for 4 days.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Questionnaire Administration
- Arm II (lavender oil) (Experimental): Patients inhale lavender essential oil via the PID once every hour starting on day 1 during their anti-cancer/chemotherapy infusions. Patients continue to inhale the lavender essential oil via the PID at least three times a day for 4 days.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Questionnaire Administration
- Arm III (ginger oil) (Experimental): Patients inhale ginger essential oil via the PID once every hour starting on day 1 during their anti-cancer/chemotherapy infusions. Patients continue to inhale the ginger essential oil via the PID at least three times a day for 4 days.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Questionnaire Administration
- Arm IV (placebo jojoba oil) (Placebo Comparator): Patients inhale placebo jojoba essential oil via the PID once every hour starting on day 1 during their anti-cancer/chemotherapy infusions. Patients continue to inhale the placebo jojoba essential oil via the PID at least three times a day for 4 days.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Aromatherapy and Essential Oils — Inhale peppermint oil
  Other Names: Aromatherapy
  Arms: Arm I (peppermint oil)
Procedure: Aromatherapy and Essential Oils — Inhale lavender oil
  Other Names: Aromatherapy
  Arms: Arm II (lavender oil)
Procedure: Aromatherapy and Essential Oils — Inhale ginger oil
  Other Names: Aromatherapy
  Arms: Arm III (ginger oil)
Procedure: Aromatherapy and Essential Oils — Inhale placebo jojoba oil
  Other Names: Aromatherapy
  Arms: Arm IV (placebo jojoba oil)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well aromatherapy essential oils work to manage anxiety and nausea in cancer patients receiving infusions in the ambulatory setting. Current drugs that are given for nausea may cause constipation and fatigue. Therefore, there is interest in exploring complementary therapies, like aromatherapy, that do not carry the same side effects. Using aromatherapy essential oils such as ginger, peppermint, and lavender, may help reduce nausea and anxiety. Some studies have shown significant reductions in nausea and anxiety among cancer patients using these oils, while other studies have had mixed results. Ginger and peppermint oils, in particular, have been associated with helping reduce nausea during chemotherapy, while lavender has shown potential benefits for anxiety. Jojoba oil will be used as a placebo for this research study. Jojoba oil is extracted from the seeds of a jojoba plant, which is a green shrub that is found in the southwestern United States). Jojoba oil is an oil which has no color or smell. Aromatherapy essential oils used through a personal inhalation device during chemotherapy may better manage anxiety and nausea in cancer patients receiving infusions in the ambulatory setting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of utilizing aromatherapy essential oils during outpatient infusions.

II. To assess satisfaction of patients receiving aromatherapy essential oils during outpatient infusions.

SECONDARY OBJECTIVES:

I. To observe whether aromatherapy essential oils (compared to placebo aromatherapy) influence an increase or decrease in nausea in patients undergoing moderate-risk and a high-risk emetogenic chemotherapy regimen.

II. To observe whether aromatherapy essential oils (compared to placebo aromatherapy) influence an increase or decrease in anxiety in patients receiving infusions in the outpatient setting.

OUTLINE: Patients are randomized to 1 of 4 arms.

ARM I: Patients inhale peppermint essential oil via the personal inhalation device (PID) once every hour starting on day 1 during their anti-cancer/chemotherapy infusions. Patients continue to inhale the peppermint essential oil via the PID at least three times a day for 4 days.

ARM II: Patients inhale lavender essential oil via the PID once every hour starting on day 1 during their anti-cancer/chemotherapy infusions. Patients continue to inhale the lavender essential oil via the PID at least three times a day for 4 days.

ARM III: Patients inhale ginger essential oil via the PID once every hour starting on day 1 during their anti-cancer/chemotherapy infusions. Patients continue to inhale the ginger essential oil via the PID at least three times a day for 4 days.

ARM IV: Patients inhale placebo jojoba essential oil via the PID once every hour starting on day 1 during their anti-cancer/chemotherapy infusions. Patients continue to inhale the placebo jojoba essential oil via the PID at least three times a day for 4 days.

After completion of study intervention, patients are followed up at day 25.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and sign a written informed consent document, and be willing to follow protocol requirements
* Ability to read and understand English for patient reported outcomes
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Willingness to comply with all study interventions of essential oil aromatherapy
* Have been on a moderate- to high-risk emetogenic chemotherapy regimen as defined by the National Comprehensive Cancer Network (NCCN) for at least 1 cycle of therapy
* At least 2 remaining infusion appointments on a moderate- to high-risk emetogenic chemotherapy regimen as defined by the NCCN
* Have nausea defined as > 3/10 with last chemotherapy infusion based on screening symptom questionnaire
* The study is open to all participants regardless of gender, race, or ethnicity

Exclusion Criteria:

* Self-reported aversion or sensitivity to lavender oil, peppermint oil, ginger oil, jojoba oil
* Uncontrolled respiratory conditions such as asthma and chronic obstructive pulmonary disease (COPD)
* Mental incapacitation (ex. stroke, brain metastasis etc.) that would cause inability to follow directions, in the opinion of the investigators
* Ongoing uncontrolled active psychiatric condition that would interfere in the conduct of the study (e.g., mood disorders, anxiety, psychosis disorders, or substance use)
* Self-reported abnormal smelling abilities (for ex: ongoing sinus infections, long covid, etc.)
* Aromatherapy use in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Participation and completion rates | At day 5 - up to 30 days post intervention
  Will consider the study feasible if >= 70% of patients are able to complete the essential oil treatment (lavender, peppermint, ginger or placebo). Completion will be defined as receiving oil treatments and submitting 4 days of at-home questionnaires as described. Will consider the study feasible if >= 50% of a patient's questionnaires are completed. Descriptive statistics will be provided to summarize all the above data.
Satisfaction of patients treated with aromatherapy essential oils | At day 5 - up to 30 days post intervention
  Will be evaluated via a post-infusion questionnaire, in order to fully understand their experience with the treatment. Will consider patients to be satisfied if >= 50% of patients answer that they are "very satisfied" or "satisfied" on their post-infusion surveys. Will also evaluate whether the patients are interested in aromatherapy essential oils for future chemotherapy infusion appointments, and their experience in the clinical trial. Descriptive statistics will be provided.

SECONDARY OUTCOMES:
Nausea scores | At day 5 - up to 30 days post intervention
  Will be evaluated between groups using data from the post-infusion questionnaire which asks, "what was the highest level of nausea that you experienced during the infusion?" as well as nausea scores from the post-infusion visual analog scale (VAS) nausea, and the Rhodes Index of Nausea, Vomiting, and Retching (INVR). Will also assess longitudinal changes in nausea scores within and between groups (VAS).
Anxiety scores I | At day 5 - up to 30 days post intervention
  Will be evaluated between groups using data from the post-infusion questionnaire which asks, "what was the highest level of anxiety that you experienced during the infusion?" as well as anxiety scores from the pre- and post-infusion Edmonton Symptom Assessment Scale (ESAS), and post-infusion VAS anxiety.
Anxiety scores II - longitudinal changes | At day 5 - up to 30 days post intervention
  Will assess longitudinal changes in anxiety scores within and between groups (VAS, State-Trait Anxiety Inventory Long Form, Edmonton Symptom Assessment System).

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lee, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California